CLINICAL TRIAL: NCT06652620
Title: A Prospective, Randomized Controlled Study on Cola Ingestion for Bolus Impaction in Patients With Esophageal Cancer
Brief Title: Cola Ingestion for Esophageal Bolus Impaction
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Kuai Le Zhao, MD, Chief physician, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ESO-Shanghai24
Record Dates: First submitted 2024-10-21; First posted 2024-10-22 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-12

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cola ingestion group (Experimental): Participants in the intervention group are instructed to consume regular Cola in an upright or sitting position after diagnosing with a complete esophageal bolus impaction.
  Interventions: Other: Cola
- Control group (No Intervention): Patients in the control group did not receive any pre-endoscopic treatment.

INTERVENTIONS:
Other: Cola — regular Coca-Cola (Coca-Cola company, Atlanta, GA) or Pesi-cola (PepsiCo, Inc.New York, NY)
  Arms: Cola ingestion group

SUMMARY:
The aim of the study is to observe whether cola ingestion can improve the 24-hour remission rate of acute esophageal impaction in patients with esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with primary esophageal lesions diagnosed by pathology, being able to consume at least a liquid diet normally before and diagnosed by a physician with acute esophageal impaction (acute esophageal impaction refers to the sudden occurrence of complete obstruction of eating within the past week)
2. Prior to enrollment, the patient did not consume carbonated beverages such as cola, or any other treatment for esophageal impaction.
3. Age ≥ 18 years old, Eastern Cooperative Oncology Group (ECOG) Performance Status score is 0-2 points.
4. The subjects voluntarily enrolled and obtained an informed consent form signed by the patient or their legal representative.

Exclusion Criteria:

1. It is known that complete esophageal obstruction is caused by tumor progression.
2. Patients who have been diagnosed with or highly suspected of having esophageal fistula through endoscopy or imaging prior to enrollment.
3. Patients with nasogastric nutrition tube and esophageal stent implantation
4. Patients who have symptoms such as coughing and are unable to drink cola, or who are at serious risk of aspiration (Glasgow Coma Scale<14 or previous history of aspiration).
5. Benign diseases such as gastroesophageal reflux, cardiac arrest, and congenital esophageal stenosis that can easily lead to foreign body impaction in the esophagus.
6. Patients with coagulation dysfunction, thrombocytopenia, or taking anticoagulant drugs that are medically considered contraindications for endoscopic examination and treatment.
7. According to the researchers' assessment, patients may not be able to cooperate with the examination and treatment, or there may be other factors that could force them to terminate the study midway, such as having other serious illnesses (including mental illnesses) that require concomitant treatment, severe abnormal laboratory test values, family or social factors, which may affect the safety of the patients or the collection of experimental data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-02-01 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
24-hour remission rate of acute esophageal impaction | The observation interval is from the diagnosis of esophageal impaction and random onset to the relief of esophageal impaction (at least allowing smooth consumption of liquid food) or the first 24-hour interval after diagnosis of esophageal impaction.
  The percentage corresponding to the ratio of the number of patients who achieved relief of esophageal impaction (including partial and complete relief) within 24 hours to the total number of patients in the group is the 24-hour relief rate.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - The Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - First People's Hospital, Jingdezhen, Jiangxi
  - Fudan University Shanghai Cancer Center, Shanghai

IPD SHARING:
Plan to Share IPD: No